CLINICAL TRIAL: NCT00767377
Title: Phase II Trial of Epirubicin, Oxaliplatin and 5-day 5-fluorouracil in Patients With Advanced and Metastatic Gastric Cancer
Brief Title: Continuous Infusion of FU Combined With Epirubicin and Oxaliplatin in Patients With A/MGC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Xiaodong Zhu, associated professor, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EOF-MGC
Record Dates: First submitted 2008-10-06; First posted 2008-10-07 (Estimated); Last update posted 2013-10-16 (Estimated); Status verified 2013-10

CONDITIONS: Gastric Cancer
Keywords: Time to Progression; Overall survival; Response rate; Quality of Live; Toxicities
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- EOF5 Group (Experimental): The regimen of 5-day Continuous infusion of FU combined with Epirubicin and Oxaliplatin will be used in the patients recruited in this trial.
  Interventions: Drug: EOF5

INTERVENTIONS:
Drug: EOF5 — epirubicin 50 mg/m2 day 1, oxaliplatin 130 mg/m2 day 1, and 5-FU 375-425 mg/m2/d day 1 through 5 continuous infusion, repeated every 3 weeks
  Other Names: treatment group

SUMMARY:
The purpose of this study is to evaluate the efficacy and tolerability of the combination of epirubicin, oxaliplatin and 5-day continuous infusional 5-fluorouracil (EOF5 regimen) in patients with unresectable advanced or metastatic gastric cancer (A/MGC). Since Mar 2011, two addition second endpoints was added to the trial, one was to compare the consistence of two types of PET Scan evaluation with routine CT Scan evaluation, the other was to search for predictor factors of clinical results ( ORR,PFS and OS) with Pharmacogenomics methods. This modification was approved by the Ethic Committee of Fudan University Cancer Hospital, and the approval number was IRB50-15-1101A.

DETAILED DESCRIPTION:
ECF regimen is considered as a reference regimen for gastric cancer in Europe. Now, no regimen has been proved to be more effective while less toxicity than ECF regimen. Oxaliplatin has demonstrated synergy with 5-FU in vitro, in vivo, and in the clinical setting in advanced colorectal cancer. It presents a better toxicity profile than cisplatin. Recently some studies used combination regimens of oxaliplatin, folinic acid, and continuous infusion 5-FU for about 44 hours (e.g FOLFOX4 ) to treat A/MGC, and yielded good response rates and median overall survival times while resulting in lower rates of grade 3-4 adverse events. Therefore, it is logical to modify ECF regimen with oxaliplatin replacing cisplatin and a short-term FU infusion replacing 21-day FU infusion. Our objective is to evaluate whether the EOF5 regimen is less toxicity while is comparable effective as ECF regimen.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed advanced or metastatic adenocarcinoma of the stomach
* ECOG performance scale ≤2
* At least one measurable lesion (larger than 10 mm in diameter by spiral CT scan)
* Adequate hepatic, renal, heart, and hematologic functions (platelets >80×109/L, neutrophil>2.0×109/L, serum creatinine ≤1.5mg/dl, total bilirubin within upper limit of normal(ULN), and serum transaminase≤2.5×the ULN)

Exclusion Criteria:

* Pregnant or lactating women
* Concurrent cancer
* History of other malignancies except cured basal cell carcinoma of skin and carcinoma in-situ of uterine cervix
* Neuropathy, brain, or leptomeningeal involvement
* Clinically relevant coronary artery disease or a history of a myocardial infarction within the last 12 months or high risk/uncontrolled arrhythmia
* Uncontrolled significant comorbid conditions and previous radiotherapy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 163 (Actual)
Dates: Start 2007-05; Primary Completion 2012-07 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Time to progression | every six weeks

SECONDARY OUTCOMES:
Toxicity | 3 weeks

OTHER OUTCOMES:
PET Scan response | 14 days
  Patients enrolled in this trial would received 18F-FLT PET SACN and 18F-FDG PET SACN before and 14 days after the first cycle chemotherapy respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Jiliang Ying, M.D, Principal Investigator — Fudan University
Locations (1):
- Fudan University Cancer Hospital, Shanghai, China